CLINICAL TRIAL: NCT07137559
Title: Expanded Access Intramuscular Injection of CELZ-201-DDT for the Treatment of Chronic Lower Back Pain
Brief Title: CELZ-201-DDT for the Treatment of Chronic Lower Back Pain
Acronym: ADAPT
Status: Available | Type: Expanded Access
Sponsor: Creative Medical Technology Holdings Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: ADAPT Expanded Access; NCT 06053242 (Other: clinicaltrials.gov)
Record Dates: First submitted 2025-08-14; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Chronic Back Pain; Degenerative Disc Disease Lumbar
Keywords: CELZ-201-DDT; Allogeneic Umbilical Cord Sub-Epithelial Cell-Derived Mesenchymal Stromal Cells; Mesenchymal Stromal Cells (MSC); Chronic Lower Back Pain; Degenerative Disc Disease (DDD); Lumbar Degeneration; Chronic Pain; Expanded Access; Single Patient IND; Emergency Use IND; Non-Emergency Use IND; Compassionate Use; Regenerative Medicine; Stem Cell Therapy
MeSH Terms: conditions — Intervertebral Disc Degeneration; Chronic Pain

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: CELZ-201-DDT — CELZ-201-DDT is administered via intramuscular injection.
  Dosing, administration, and follow-up will be determined by the treating physician in accordance with the EA authorization and medical judgment. Safety monitoring will be performed during and after treatment, and all serious adverse events will be reported to the FDA and IRB per applicable regulations.

SUMMARY:
CELZ-201-DDT is an investigational (experimental) cell therapy currently being studied for people with degenerative disc disease who have chronic lower back pain.

DETAILED DESCRIPTION:
Expanded Access to CELZ-201-DDT (Allogeneic Umbilical Cord Sub-Epithelial Cell-Derived Mesenchymal Stromal Cells) is available for individual patients with serious or life-threatening chronic lower back pain due to degenerative disc disease (DDD) who have no comparable or satisfactory alternative therapy options.

Requests will be considered on a case-by-case basis under a single-patient IND in coordination with the U.S. Food and Drug Administration (FDA) and an Institutional Review Board (IRB).

For non-emergency requests, the treating physician must submit FDA Form 3926 and obtain FDA authorization before initiating treatment.

For emergency use, treatment may begin without prior FDA authorization if criteria for emergency use are met; the physician must notify the FDA within 5 working days after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of chronic lower back pain due to degenerative disc disease.
* No comparable or satisfactory alternative therapy available. Unable to participate in the ongoing CELZ-201-DDT clinical trial. Informed consent provided.

Exclusion Criteria:

* Any medical condition that poses an unacceptable risk or would interfere with treatment safety or evaluation.
* Known hypersensitivity to any component of the investigational product.

How to Request Access:

* Contact the Expanded Access Coordinator to confirm eligibility and discuss feasibility.
* Complete and submit FDA Form 3926 to the appropriate FDA review division.
* Obtain IRB review (may be expedited or post-treatment for emergency use). Coordinate drug shipment and treatment schedule.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult